CLINICAL TRIAL: NCT00280397
Title: An Open Label Phase I Dose Escalation Study of E7080 Administered to Patients With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E7080-J081-103
Record Dates: First submitted 2006-01-20; First posted 2006-01-23 (Estimated); Results first posted 2015-03-06 (Estimated); Last update posted 2016-10-07 (Estimated); Status verified 2016-08

CONDITIONS: Cancer: Solid Tumors
Keywords: Cancer, solid tumors
MeSH Terms: conditions — Neoplasms | interventions — lenvatinib

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: E7080

INTERVENTIONS:
Drug: E7080 — E7080 is administered orally twice a day for 2 weeks to patients with solid tumors that are resistant to approved conventional therapies or for which no appropriate treatment is available.

SUMMARY:
The purpose of this study is to determine the maximum tolerable dose (MTD) and the related effects of E7080 administered to patients with solid tumors that are resistant to approved existing anti-tumor therapies, or for which no appropriate treatment is available.

ELIGIBILITY:
Inclusion criteria:

1. Patients who have histologically and/or cytologically confirmed solid tumors requiring treatment.
2. Patients with solid tumors which are resistant to approved conventional anti-tumor therapies, or for which no appropriate treatment is available.
3. Patients who had completed all previous treatments (including surgery and radiotherapy) and supportive care (such as transfusion of blood, blood components and granulocyte colony-stimulating factor [G-CSF] treatment) at least 4 weeks before registration, and no sign or symptom of acute toxicity occurred in previous treatments.
4. Patients 20 years or older and less than 75 years of age at the time of registration.
5. Patients with 0 or 1 Performance Status (PS) established by Eastern Cooperative Oncology Group (ECOG.)
6. Patients who can stay in hospital for more than 1 cycle of treatment.
7. Patients who are expected to survive for more than 3 months from the start of study drug administration.
8. Patients who have provided written informed consent for the participation in the study.

Exclusion criteria:

1. Patients with clinical symptoms due to brain metastases requiring treatment.
2. Patients who have any of the following laboratory test findings:

   1. Hemoglobin less than 9.0 g/dL
   2. Neutrophil count less than 1.5 x 10 9/L
   3. Platelet count less than 100 x 10 9/L
   4. Serum bilirubin greater than 1.5 mg/dL
   5. AST, ALT greater than 100 IU/L
   6. Serum creatinine greater than 1.5 mg/dL or creatinine clearance less than 50 mL/minute
3. Patients with positive reaction for human immunodeficiency virus (HIV) or hepatitis virus C (HCV) antibody or hepatitis B virus surface (HBs) antigen, or patients with untreated serious infections.
4. Patients with clinically significant cardiac disorders or unstable ischemic heart diseases including myocardial infarction within six months before the registration for the study.
5. Patients with marked Baseline prolongation of QT/QTc interval (QTc interval greater than 450 msec for males or greater than 470 msec for females) using the Fridericia method for QTc analysis.
6. Patients with hemorrhagic or thrombotic diseases or who are using therapeutic doses of anticoagulants such as aspirin, warfarin, or ticlopidine.
7. Patients who are diagnosed with hypertension (defined as repeatedly measured blood pressure = 160/90 mmHg) at Screening, irrespective of use of antihypertensive drugs.
8. Patients who have proteinuria greater than 1 on bedside testing.
9. Patients who have history of insufficient gastrointestinal absorption, or patients who received gastric or intestinal anastomoses within 4 weeks before registration.
10. Patients who have history of alcoholism, drug addiction or mental or physical disorders, which, in the investigators opinion, may impair study compliance.
11. Patients who received any investigational drug within 30 days before the registration of the study.
12. Patients who received CYP3A4 inhibitors including itraconazole, erythromycin, clarithromycin, diltiazem or verapamil during screening and who have to use these drugs during the study.
13. Pregnant or nursing patients (all female patients with pregnancy potential must have negative pregnancy test performed before registration, and post-menopausal women must be amenorrheic for at least 12 months.) Female patients must use appropriate contraception.
14. Fertile male patients who refuse to use contraception, or whose female partners are not using appropriate contraception.
15. Patients who are judged by the investigator to be inappropriate for the study.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2006-01; Primary Completion 2008-09 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Akihiko Tsuruoka, Study Director — Eisai Co., Ltd.
Locations (1):
- Tokyo, Tokyo, Japan

REFERENCES:
- [Derived] Koyama N, Saito K, Nishioka Y, Yusa W, Yamamoto N, Yamada Y, Nokihara H, Koizumi F, Nishio K, Tamura T. Pharmacodynamic change in plasma angiogenic proteins: a dose-escalation phase 1 study of the multi-kinase inhibitor lenvatinib. BMC Cancer. 2014 Jul 21;14:530. doi: 10.1186/1471-2407-14-530. PMID 25047123
- [Derived] Yamada K, Yamamoto N, Yamada Y, Nokihara H, Fujiwara Y, Hirata T, Koizumi F, Nishio K, Koyama N, Tamura T. Phase I dose-escalation study and biomarker analysis of E7080 in patients with advanced solid tumors. Clin Cancer Res. 2011 Apr 15;17(8):2528-37. doi: 10.1158/1078-0432.CCR-10-2638. Epub 2011 Mar 3. PMID 21372218

RESULTS

PARTICIPANT FLOW:
Groups:
- E7080 Group: E7080 is administered orally twice a day for 2 weeks to patients with solid tumors that are resistant to approved conventional therapies or for which no appropriate treatment is available.
Period: Overall Study
Arm/Group | E7080 Group
Started | 27
Completed | 26
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | E7080 Group
Number analyzed (Participants) | 27
Age, Continuous [Mean (Standard Deviation); unit: Years] | 50.7 (11.1)
Sex/Gender, Customized [Number; unit: Participants]
  Male | 10
  Female | 17

OUTCOME MEASURES:

1. Secondary Outcome: To Elucidate the Pharmacokinetic Profile of E7080
Time Frame: Every 3 weeks
Reporting Status: Not Posted

2. Primary Outcome: Maximum Tolerable Dose (MTD) of E7080 Repeatedly Administered Twice a Day
Description: The MTD was defined as the highest dose at which no dose limiting toxicity (DLT) was experienced by the first 3 patients in that cohort, or the dose at which a DLT was experienced by no more than 1 of 6 patients evaluable for toxicity.
Time Frame: up to 4 weeks
Population: Registered participants were included in the tolerability analysis set with the exception of the ineligible participants, participants with a treatment compliance rate of less than 75%, and participants who discontinued the study for reasons other than occurrence of DLT. However, cases of DLT shall be included in analyses.
Measure: Number; unit: mg BID
Arm/Group | E7080 Group
Number analyzed (Participants) | 26
mg BID | 13

3. Secondary Outcome: Number of Participants With Adverse Events / Serious Adverse Events
Description: Treatment emergent adverse events (AEs) and serious adverse events (SAEs) were evaluated.
Time Frame: Until tumor progression, unacceptable toxicity, or withdrawal due to other reasons.
Population: All participants who received at least one E7080 dose and had evaluable data were included in the safety analyses.
Measure: Number; unit: Participants
Arm/Group | E7080 Group
Number analyzed (Participants) | 27
Participants | 27

4. Primary Outcome: DLT of E7080 Repeatedly Administered Twice a Day
Description: DLTs were defined as grade 3 or more platelet count decrease, grade 4 neutropenia, any grade 3 or more nonhematologic toxicity (with exceptions of grade 4 hypertension not controlled by any antihypertensive drugs and grade greater than or equal to 3 vomiting and diarrhea not controlled by antiemetic or antidiarrheal drugs), and failure to administer more than 75% of the planned doses of E7080 during the same cycle due to toxicity.
Time Frame: up to 4 weeks
Population: as for outcome 2
Measure: Number; unit: Participants with DLT
Groups:
- E7080 - 16 mg Group; E7080 - 20 mg Group: E7080 is administered orally twice a day for 2 weeks to patients with solid tumors that are resistant to approved conventional therapies or for which no appropriate treatment is available.
Arm/Group | E7080 - 16 mg Group | E7080 - 20 mg Group
Number analyzed (Participants) | 3 | 3
Participants with DLT | 1 | 2

5. Secondary Outcome: Determine the Clinical Dose for Phase II Study Based on Safety and Pharmacokinetic Profile
Time Frame: Every 3 weeks
Reporting Status: Not Posted

6. Secondary Outcome: Evaluate the Anti-tumor Activity of E7080
Time Frame: Every 3 weeks
Reporting Status: Not Posted

7. Secondary Outcome: To Make Exploratory Analyses of Pharmacodynamic Markers
Time Frame: Every 3 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Until tumor progression, unacceptable toxicity, or withdrawal due to other reasons.
Description: All participants who received at least one E7080 dose and had evaluable data were included in the safety analyses. Treatment emergent adverse events (AEs) and serious adverse events (SAEs) were evaluated.
Arm/Group | E7080 Group
Serious Adverse Events (participants affected / at risk) | 7/27
Other Adverse Events (participants affected / at risk) | 27/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | E7080 Group (N=27)
Hypertension (Vascular disorders) | 2
Postrenal failure (Renal and urinary disorders) | 1
Haemorrhage (Vascular disorders) | 1
Pneumonia (Infections and infestations) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Platelet count decreased (Investigations) | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | E7080 Group (N=27)
Anaemia (Blood and lymphatic system disorders) | 6
Sinus bradycardia (Cardiac disorders) | 2
Eyelid oedema (Eye disorders) | 3
Abdominal pain (Gastrointestinal disorders) | 2
Abdominal pain upper (Gastrointestinal disorders) | 5
Constipation (Gastrointestinal disorders) | 7
Diarrhoea (Gastrointestinal disorders) | 15
Gingival bleeding (Gastrointestinal disorders) | 2
Gingivitis (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 12
Stomach discomfort (Gastrointestinal disorders) | 2
Stomatitis (Gastrointestinal disorders) | 5
Vomiting (Gastrointestinal disorders) | 8
Chest pain (General disorders) | 2
Face oedema (General disorders) | 4
Fatigue (General disorders) | 19
Malaise (General disorders) | 2
Oedema (General disorders) | 2
Oedema peripheral (General disorders) | 10
Pyrexia (General disorders) | 3
Nasopharyngitis (Infections and infestations) | 9
Tonsillitis (Infections and infestations) | 2
Procedural pain (Injury, poisoning and procedural complications) | 3
Alanine aminotransferase increased (Investigations) | 15
Aspartate aminotransferase increased (Investigations) | 17
Blood albumin decreased (Investigations) | 13
Blood alkaline phosphatase increased (Investigations) | 13
Blood bilirubin increased (Investigations) | 4
Blood calcium decreased (Investigations) | 2
Blood cholesterol increased (Investigations) | 5
Blood creatine phosphokinase increased (Investigations) | 3
Blood creatinine increased (Investigations) | 7
Blood fibrinogen increased (Investigations) | 10
Blood lactate dehydrogenase increased (Investigations) | 14
Blood potassium increased (Investigations) | 2
Blood sodium decreased (Investigations) | 4
Blood thyroid stimulating hormone increased (Investigations) | 7
Blood triglycerides increased (Investigations) | 2
Blood urea increased (Investigations) | 7
Blood uric acid increased (Investigations) | 4
Blood urine present (Investigations) | 20
C-reactive protein increased (Investigations) | 2
Electrocardiogram T wave amplitude decreased (Investigations) | 3
Gamma-glutamyltransferase increased (Investigations) | 11
Glucose urine present (Investigations) | 3
Haemoglobin decreased (Investigations) | 2
Leucine aminopeptidase increased (Investigations) | 4
Lymphocyte count decreased (Investigations) | 2
Neutrophil count decreased (Investigations) | 5
Neutrophil count increased (Investigations) | 2
Platelet count decreased (Investigations) | 10
Platelet count increased (Investigations) | 2
Protein total decreased (Investigations) | 9
Protein urine present (Investigations) | 17
Red blood cell count decreased (Investigations) | 3
Weight decreased (Investigations) | 4
Weight increased (Investigations) | 2
White blood cell count decreased (Investigations) | 7
White blood cell count increased (Investigations) | 3
Anorexia (Metabolism and nutrition disorders) | 12
Hypercholesterolaemia (Metabolism and nutrition disorders) | 2
Hyperlipidaemia (Metabolism and nutrition disorders) | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Dizziness (Nervous system disorders) | 6
Headache (Nervous system disorders) | 17
Insomnia (Psychiatric disorders) | 2
Haematuria (Renal and urinary disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 3
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 2
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 5
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 4
Rash (Skin and subcutaneous tissue disorders) | 5
Hot flush (Vascular disorders) | 4
Hypertension (Vascular disorders) | 17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Other disclosure agreement that restricts the right of the PI to discuss or publish trial results after the trial is completed.